CLINICAL TRIAL: NCT05894200
Title: Effectiveness and Retention of Pit and Fissure Sealants in Rural Setup: A School-based Clinical Trial in Nepal
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Kathmandu University School of Medical Sciences (Other)
Collaborators: University Grants Commission (Other)
Responsible Party: Principal Investigator, Dilip Prajapati, Assistant professor, Kathmandu University School of Medical Sciences
Other Study IDs: 66/23
Record Dates: First submitted 2023-05-29; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Dental Caries Pit and Fissure; Oral Disease
Keywords: Nepal; Oral health; Dental
MeSH Terms: conditions — Mouth Diseases | interventions — Pit and Fissure Sealants; silver diamine fluoride

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Glass Ionomer cement pit and fissure sealant, Silver Diamine Fluoride — GC Fuji 7, e-SDF

SUMMARY:
The program titled "Campus to Community: breaking the barrier in oral health education and dental care" is uniquely designed program to link University (Kathmandu University School of Medical Sciences) to community (Sanghutar, Ramechhap). Dhulikhel Hospital, Kathmandu University Teaching Hospital has established a model dental clinic in the premises of Him Ganga Secondary School, Shangutar which is operated by council registered Dentist and dental hygienist. The objective of this study is to assess oral health condition of the children aged 6-15 years of the school followed by application of pit and fissure sealant (PFS) in non-carious permanent molar and Silver diamine fluoride (SDF) in carious permanent teeth. Data will be recorded according to the WHO Oral health assessment form for children, 2013 by a calibrated dentist from Dhulikhel Hospital and retention of PFS and efficacy of SDF application will be followed up after 6 months by the same investigators. The program is proposed with the expectation that proper oral hygiene prevention program combined with preventive procedures like pit and fissure sealant and SDF can reduce the burden of oral diseases in rural setup.

DETAILED DESCRIPTION:
World Health Organization reported that untreated caries in permanent teeth is the most prevalent condition, affecting 3.5 billion people globally, which seems more aggressive in developing countries. Such untreated dental caries in permanent teeth is the most common health condition according to the global burden of disease 2019 which can be largely preventable and school based preventive program are the most effective one to overcome such problems. Acute or unplanned dental care accounted loss of 34 million school hours annually compared to children with very good oral health. Silver diamine fluoride is safe and effective alternative treatment for the children which can improve oral health outcomes for community members especially for individuals from low socioeconomic settings and can transform the concept of community dental caries program. pit and fissure sealants is very effective tool for caries prevention on an individual basis or as part of a public health measure for at - risk populations which can be applied both primary and secondary level of prevention. However in developing and underdeveloped countries, because of the lack of this preventive measure, every year children develop dental caries, pulpitis and ultimately extraction of permanent teeth which could otherwise be saved.

Methodology: Screening will be done in the school premises by the expert dentist from Kathmandu University School of Medical Science with sterilized Dental kit and head lamp taking universal precautions. Participants will be segregated according to class and respective class teachers will help them in screening accordingly. Both verbal and written consent will be taken from students, respective class teachers and parents if available.

World health organization, Oral Health Assessment form for Children, 2013 will be used to collect oral health data which includes demographic details, dentition status, gingival status, enamel fluorosis, Dental trauma, oral mucosal lesions, intervention urgency and dento-facial anomalies. After recording the data, Investigator will make a treatment plan and segregate the students according to the need for Silver diamine fluoride application, GIC pit and fissure sealant application or oral urgency treatment which will be coordinated by the available volunteers. All the students who participated in this study will be provided with fluoridated toothpaste and brush.

Pit and fissure sealant application: Deep pit and fissure will be identified and plaque removal is done with the toothbrush provided, conditioning will be done by conditioner liquid available with GIC pit and fissure sealant. Tooth surface will be cleaned with three-way syringe available in dental chair, Isolation will be maintained with cotton roll and sealant will be evaluated and occlusal bite will be registered. Students will be informed about post-restoration instructions in verbal and printed form of instruction will be given to individuals.

ELIGIBILITY:
Inclusion Criteria:

* All the students from the school who is willing to participate in this study aged between 6-15 years old

Exclusion Criteria:

* Students who is not willing to participate or not permitted from parents

Ages: 6 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: Purposive sampling technique used among school children from Him Ganga secondary School, Shangutar, Ramechhap , Nepal
Sampling Method: Non-Probability Sample
Enrollment: 377 (Estimated)
Dates: Start 2023-08-10 (Estimated); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-25 (Estimated)

PRIMARY OUTCOMES:
Effectiveness and Retention of Pit and Fissure Sealants in Rural Setup: A School-based Clinical Trial in Nepal | one year
  Effectiveness of pit and fissure sealant in permanent molars, change from baseline in retention of the sealant at six months

SECONDARY OUTCOMES:
Effectiveness of silver diamine fluoride in caries prevention and arrest: An observational rural school based study | one year
  Rate of arrested dental caries on permanent first molars with SDF application within one year followup

CONTACTS AND LOCATIONS:
Overall Officials: Dashrath Kafle, MDS, Study Director — KUSMS
Locations (1):
- Kathmandu University, Kavre, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Undecided
if needed , will share IPD

REFERENCES:
- [Result] Beauchamp J, Caufield PW, Crall JJ, Donly K, Feigal R, Gooch B, Ismail A, Kohn W, Siegal M, Simonsen R; American Dental Association Council on Scientific Affairs. Evidence-based clinical recommendations for the use of pit-and-fissure sealants: a report of the American Dental Association Council on Scientific Affairs. J Am Dent Assoc. 2008 Mar;139(3):257-68. doi: 10.14219/jada.archive.2008.0155. PMID 18310730
- [Result] Alkhodairi A, Alseweed M, Alwashmi S, Elmoazen RA. Clinical Evaluation of the Retention of Resin and Glass Ionomer Sealants Applied as a Part of School-Based Caries Prevention Program. Open Access Maced J Med Sci. 2019 Dec 13;7(23):4127-4130. doi: 10.3889/oamjms.2019.869. eCollection 2019 Dec 15. PMID 32165964
- [Result] Bridge G, Martel AS, Lomazzi M. Silver Diamine Fluoride: Transforming Community Dental Caries Program. Int Dent J. 2021 Dec;71(6):458-461. doi: 10.1016/j.identj.2020.12.017. Epub 2021 Feb 27. PMID 33653594
- See also: Central bureau of statistic, Government of Nepal Census 2021 — http://citypopulation.de/en/nepal/admin/bagmati/21ramechhap/
- See also: World Health organization. Oralhealth survey fifth edition — https://www.who.int/news-room/fact-sheets/detail/oral-health